CLINICAL TRIAL: NCT00557154
Title: Ultrasound Assisted Peripheral Venous Access in Young Children: A Pilot and Feasibility Randomized Controlled Trial
Brief Title: Ultrasound Assisted Peripheral Venous Access in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Children's Miracle Network (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200210274; S-9400847-018LA (Other: Other)
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2007-11

CONDITIONS: Catheterization, Peripheral
Keywords: Pediatrics; Venous access; Emergency
MeSH Terms: conditions — Emergencies | interventions — Ultrasonography; Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Ultrasound used to visualize peripheral venous anatomy. This guides subsequent attempts at venipuncture.
  Interventions: Device: ultrasound
- 2 (Active Comparator): Routine venipuncture using standard methods.
  Interventions: Device: standard technique for venipuncture

INTERVENTIONS:
Device: ultrasound — ultrasound used to identify target vein
  Arms: 1
Device: standard technique for venipuncture — routine equipment
  Arms: 2

SUMMARY:
The purpose of this study is to learn how the use of ultrasound helps with the placement of an intravenous (i.v.) catheter in young children.

DETAILED DESCRIPTION:
In an academic pediatric Emergency Depratment (ED), we performed a randomized clinical trial of children < 7 years of age, who required i.v. access and who had failed the first i.v. attempt. We randomized patients to either continued standard i.v. attempts or ultrasound-assisted attempts. Clinicians involved in the study received one hour of training in ultrasound localization of peripheral veins. In the ultrasound group, vein localization was performed by an ED physician who marked the skin overlying the target vessel. Intravenous cannulation attempts were then immediately performed by a pediatric ED nurse who relied on the skin mark for vessel location. We allowed for technique cross-over after two failed i.v. attempts. We recorded success rate and location of access attempts.

ELIGIBILITY:
Inclusion Criteria:

* Less than 7 years of age
* Emergency Department patients
* Parents available for consent

Exclusion Criteria:

* Critical illness

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2003-08; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
venous visualization (with ultrasound) and venipuncture success rate | one year

SECONDARY OUTCOMES:
Anticipated difficulty of venipuncture (rated on visual analog scale) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Aaron E Bair, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States